CLINICAL TRIAL: NCT00396370
Title: Phase I Studies of the Safety and Immunogenicity of Primary and Secondary BCG Vaccination Delivered Intradermally, Orally and by Combined Routes of Administration in Healthy and Previously Immunologically Naïve Volunteers
Brief Title: BCG Vaccination Delivered Intradermally, Orally and by Combined Routes
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 01-351
Record Dates: First submitted 2006-11-03; First posted 2006-11-06 (Estimated); Last update posted 2019-11-12 (Actual); Status verified 2012-10-26

CONDITIONS: Tuberculosis
Keywords: Bacillus Calmette-Guérin; parent protocol; tuberculosis
MeSH Terms: conditions — Tuberculosis

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (7):
- Group A: BCG ID/Placebo PO; Placebo ID/Placebo PO (Experimental): Primary vaccination: BCG ID (Danish)/Placebo PO; secondary vaccination (1 year later): Placebo ID/Placebo PO.
  Interventions: Biological: BCG strain Danish; Other: Placebo
- Group B: BCG ID/Placebo PO; BCG ID/Placebo PO (Experimental): Primary vaccination: BCG ID (Danish)/Placebo PO; secondary vaccination (1 year later): BCG ID (Danish)/Placebo PO.
  Interventions: Biological: BCG strain Danish; Other: Placebo
- Group C: Placebo ID/BCG PO; Placebo ID/Placebo PO (Experimental): Primary vaccination: Placebo ID/BCG PO (Danish); secondary vaccination (1 year later): Placebo ID/Placebo PO.
  Interventions: Biological: BCG strain Danish; Other: Placebo
- Group D: Placebo ID/BCG PO; Placebo ID/BCG PO (Experimental): Primary vaccination: Placebo ID/BCG PO (Danish); secondary vaccination (1 year later): Placebo ID/BCG PO (Danish).
  Interventions: Biological: BCG strain Danish; Other: Placebo
- Group E: BCG ID/BCG PO; Placebo ID/Placebo PO (Experimental): Primary vaccination: BCG ID (Danish)/BCG PO (Danish); secondary vaccination (1 year later): Placebo ID/Placebo PO.
  Interventions: Biological: BCG strain Danish; Other: Placebo
- Group F: BCG ID/BCG PO; BCG ID/BCG PO (Experimental): Primary vaccination: BCG ID (Danish)/BCG PO (Danish); secondary vaccination (1 year later): BCG ID (Danish)/BCG PO (Danish).
  Interventions: Biological: BCG strain Danish
- Group G: Connaught strain BCG ID (Experimental): Primary vaccination: Connaught strain BCG ID; secondary vaccination (1 year later): none.
  Interventions: Biological: BCG strain Connaught

INTERVENTIONS:
Biological: BCG strain Connaught — Connaught strain Bacillus Calmette-Guerin (BCG), 8-32 x 10^5 CFU vaccine for intradermal administration.
  Arms: Group G: Connaught strain BCG ID
Biological: BCG strain Danish — Bacillus Calmette-Guerin (BCG) strain Danish from the Statens Serum Institute (SSI BCG). 1.2 X 10^8 colony-forming units (CFU) oral (PO) in 60 mililiters phosphate buffered saline (PBS).
  Arms: Group C: Placebo ID/BCG PO; Placebo ID/Placebo PO; Group D: Placebo ID/BCG PO; Placebo ID/BCG PO; Group E: BCG ID/BCG PO; Placebo ID/Placebo PO; Group F: BCG ID/BCG PO; BCG ID/BCG PO
Biological: BCG strain Danish — Bacillus Calmette-Guerin (BCG) strain Danish from the Statens Serum Institute (SSI BCG). 2-8 X 10^5 colony-forming units (CFU) intradermal in 100 microliters diluent.
  Arms: Group A: BCG ID/Placebo PO; Placebo ID/Placebo PO; Group B: BCG ID/Placebo PO; BCG ID/Placebo PO; Group E: BCG ID/BCG PO; Placebo ID/Placebo PO; Group F: BCG ID/BCG PO; BCG ID/BCG PO
Other: Placebo — 0.1 mL of sterile Sauton medium for intradermal administration.
  Arms: Group A: BCG ID/Placebo PO; Placebo ID/Placebo PO; Group C: Placebo ID/BCG PO; Placebo ID/Placebo PO; Group D: Placebo ID/BCG PO; Placebo ID/BCG PO; Group E: BCG ID/BCG PO; Placebo ID/Placebo PO
Other: Placebo — 60 mL of sterile phosphate buffered saline (PBS) for oral administration.
  Arms: Group A: BCG ID/Placebo PO; Placebo ID/Placebo PO; Group B: BCG ID/Placebo PO; BCG ID/Placebo PO; Group C: Placebo ID/BCG PO; Placebo ID/Placebo PO; Group E: BCG ID/BCG PO; Placebo ID/Placebo PO

SUMMARY:
This study will assess the safety of a Bacillus Calmette-Guérin (BCG) vaccine against tuberculosis (TB) and will evaluate if giving the vaccine by mouth, injection, or by both methods produces greater results. BCG vaccine and/or placebo (substance containing no medication) will be given by mouth and/or by injection into the skin. This study, conducted at Saint Louis University, will enroll 60 (up to 80) healthy volunteers, 18-40 years old, who are negative for a TB test (QuantiFERON®-Gold) and human immunodeficiency virus (HIV). Study procedures will include a physical exam; review of TB exposure history and medical history; collection of multiple samples of blood, urine, stool, tears, and nose fluid; and skin and blood tests for TB. Volunteers may participate for about 24 months.

DETAILED DESCRIPTION:
Vaccination with Bacillus Calmette-Guérin (BCG) is used as part of tuberculosis (TB) control strategies in most of the world outside of the United States and constitutes the most widely implemented vaccination strategy worldwide. However, despite widespread use of BCG, TB remains a leading infectious cause of death worldwide and it is estimated that one-third of the world's population is chronically and asymptomatically (latently) infected with Mycobacterium tuberculosis (Mtb), the causative agent of TB. This is a phase I, single-center, randomized, vaccine trial including six double-blind, placebo-controlled groups and one open-label group. Approximately 68 (up to 80) healthy male and female subjects 18-40 years old, inclusive, who are negative for QuantiFERON®-TB Gold and human immunodeficiency virus will be enrolled. The expected total duration of the volunteer enrollment, vaccination, and follow-up (volunteer participation) for this study is 30 months. All volunteers are expected to be enrolled over a period of 9 months and on study for 24 months. Detailed immune studies with frozen samples will be expected to continue after collection of all samples and after the protocol has been completed. Eligibility will be determined by volunteer's health at prescreening and eligible subjects will give study specific main study informed consent for enrollment in the study. Subjects randomized to Groups A-F will receive, at Day 0 and 1 year later, BCG intradermally, orally, or by both routes. PBS (PO) and Sauton medium (injectable) placebo will be used to blind the study. Subjects randomized to Group G will receive BCG intradermally at Day 0 only. The primary study objectives are the assessment of the safety of combined and individual intradermal (ID) and oral (PO) vaccination with Statens Serum Institut (SSI) BCG in healthy, immunologically naïve volunteers; comparisons of mycobacteria-specific interferon-gamma responses and mucosal immunoglobulin-A induced by SSI BCG vaccination given intradermally, orally and by both routes combined; and comparison of safety and immunogenicity of Danish and Connaught BCG given intradermally. The secondary study objectives are the assessment of purified protein derivative skin test responses as an indication of cutaneous T cell trafficking after vaccination with SSI BCG; and quantitation of BCG replication in Sanofi Pasteur ID BCG ulcerative lesions after ID BCG vaccination. The exploratory study objectives are comparisons of intracellular killing activity induced by SSI BCG vaccination given intradermally, orally, and by both routes combined; and characterization of mycobacteria-specific T cells induced intradermally, orally, or both routes by vaccination with SSI BCG using dendritic cells as antigen-presenting cells and stored peripheral blood mononuclear cells as a source for matched T cells collected before and after vaccination. Parent protocol to sub-study 12-0110 and 10-0026.

ELIGIBILITY:
Inclusion Criteria:

-Demonstrate adequate understanding of the study and its requirements for participation, as demonstrated by the responses on a written assessment tool, discussions with the study staff, and ability to provide written informed consent to participate in the research study. -Be 18 to 40 years of age, inclusive. -Be available for a total of up to 36 months of follow-up (for those volunteers interested in the leukapheresis procedure). -Weigh at least 110 pounds. -Male or female. Females must not be pregnant, as determined by negative serum pregnancy test at screening, have a negative urine pregnancy test on the day of vaccination, and must be non-lactating. -Women will use an effective method of contraception (licensed hormonal treatment, monogamous relationship with vasectomized partner, surgical sterilization, barrier method such as diaphragm or condom with contraceptive foam or total abstinence) for 30 days prior to immunization and for the 2-year period of study follow-up. -Be in good health as judged by a physician on the basis of reported medical history and physical examination including blood pressure (BP) and respiratory evaluation. -Have a negative human immunodeficiency virus (HIV)-1 enzyme-linked immunosorbent assay (ELISA) test. -Have negative serology tests for hepatitis B surface antigen and hepatitis C virus antibody. -Have a negative QuantiFERON®-tuberculosis (TB) Gold test, defined as early secretory antigenic target (ESAT)-6 response minus nil response < 0.35 IU/ml, CFP-10 response minus nil response <0.35 IU/ml, nil response less than or equal to 0.7 IU/ml, and mitogen response greater than or equal to 0.5 IU/ml. -Have clinical hematologic and chemistry laboratory results within normal values for age and gender. For creatinine and aspartate aminotransferase (AST) levels, the applicable cut-offs for determination of normal are the upper limits of normal only, as there is no clinical significance associated with results below the lower limits of normal for these laboratory values. -Have a urine dipstick test negative for glucose and </=1 plus for protein. -Access to a telephone.

Exclusion Criteria:

-Have a history of suspected or confirmed active tuberculosis (symptoms may include recurrent fever, fatigue, night sweats, weight loss, oral ulcers, diarrhea, nausea or vomiting, bleeding). -Have any systemic symptoms including fever, malaise, fatigue, chills, night sweats, weight loss, nausea, vomiting or bleeding, diarrhea, abdominal pain, rhinorrhea, cough, wheezing, or shortness of breath within 72 hr before vaccination or signs of mucosal ulceration, lymphadenitis, gastrointestinal, or pulmonary disease by physical examination on day of vaccination. -Note: Systemic symptoms occurring prior to secondary vaccination will result in the secondary vaccination being delayed until at least 72 hr after resolution of any of these symptoms that were not considered indicative of active tuberculosis (TB). -Have lymphadenopathy, hepatosplenomegaly, or other abnormalities on physical examination. -Have oropharyngeal or skin ulceration, or history of chronic/recurrent peptic ulcer disease or gastritis. -Note: Self-limited ulceration at intradermal (ID) vaccination site healing within 3 months or other mild to moderate complaints lasting less than 1-2 weeks, as documented in the memory aids (used for 2 weeks after each vaccination) or other source documents used to capture results of clinical assessments at any time point during the trial, will not be reasons to exclude a volunteer from receiving the secondary vaccination. -History of any significant acute or chronic medical conditions including, but not limited to, disorders of the liver, kidney, lung, heart, or nervous system, or other metabolic or autoimmune/inflammatory conditions. -Have any history of scarring badly or keloid formation. -Have identifiable intermediate or high-risk behavior for HIV infection (defined as having had unprotected intercourse with multiple partners in the past year prior to enrollment, including men having sex with men). -Lives with someone with HIV, acquired immune deficiency syndrome (AIDS) or active cancer. -Have chronic administration (defined as more than 14 days) of immunosuppressants or other immune-modifying drugs within 6 months prior to the vaccine dose. (For corticosteroids, this will mean prednisone, or equivalent, greater than or equal to 0.5 mg/kg/day. Inhaled and topical steroids are allowed.) -Have a history of smoking, alcoholism requiring medical attention, substance abuse, and/or intravenous drug use within the past 1 year prior to enrollment in the study. -Has a history or physical findings to suggest asthma or any chronic pulmonary condition. -Has a history of epilepsy. -Has a pacemaker or implantable cardiac devices. -Has a prosthetic valve. -Has a history of bleeding disorder. -Known allergy to any vaccine components. -Is currently taking anticoagulant or anti-platelet drugs and/or insulin. -Is currently under a physician's care for asthma or any chronic pulmonary condition. -Received blood products or immunoglobulin within 6 months of the first vaccination. -Vaccinated previously with Bacillus Calmette-Guérin (BCG) at study entry. -Received live attenuated vaccines within 4 weeks of vaccination. -Received inactivated vaccines within 2 weeks of vaccination. (Medically indicated inactivated vaccines should be given at least 2 weeks away from BCG immunization, or any sampling time point after vaccination.) -Participated in another research study that includes receiving an experimental agent or drug 30 days prior to vaccination. -Have a history of the use of a systemic antibiotic within the 14 days prior to vaccination or planned use of a systemic antibiotic during this study. -Have any medical, psychiatric, occupa tional, or behavioral problems that make it unlikely the volunteer will comply with the protocol as determined by the principal investigator (PI). -Be a health care provider at the highest risk of acquiring Mycobacterium tuberculosis (Mtb) infection, such as pulmonologists performing bronchoscopies on TB patients.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 69 (Actual)
Dates: Start 2008-12-02 (Actual); Primary Completion 2012-07-23 (Actual); Study Completion 2012-07-23 (Actual)

PRIMARY OUTCOMES:
Immunogenicity: post-vaccination increases in mycobacteria-specific Th1 responses measured by both 7 day whole blood interferon (IFN)-gamma secretion and overnight IFN-gamma enzyme linked immunospot (ELISPOT) assays. | Harvested immediately before primary vaccination, and 1 week, 2, 6, and 12 months after primary vaccination, and 1 week, 2, 6, and 12 months after secondary vaccination.
Immunogenicity: post-vaccination mycobacteria-specific secretory immunoglobulin A (IgA) responses measured by enzyme-linked immunosorbent assay (ELISA). | Harvested immediately before primary vaccination, and 1 week, 2, 6, and 12 months after primary vaccination, and 1 week, 2, 6, and 12 months after secondary vaccination.
Microbiologic: variability of Bacillus Calmette-Guérin (BCG) replication in intradermal (ID) ulcerative lesions in Group G. | Days 7, 13-15, 20-22, 27-29, 34-36 and 41-43, and 2 months following ID BCG vaccination.
Safety: incidence of adverse events. | Solicited symptoms Days 0-14 after each vaccination, unsolicited adverse events collected for 2 months after each vaccination, serious adverse events collected through 12 months after the last vaccination.

SECONDARY OUTCOMES:
Immunogenicity: presence or absence of cutaneous T cell trafficking, as indicated by purified protein derivative (PPD) skin test responses as an indication of cutaneous T cell trafficking after vaccination with SSI BCG. | Assessed in the study 2 years after primary vaccination with SSI BCG.
Immunogenicity: proportion of subjects in each treatment group achieving an immunologically significant increase in primary endpoint Mtb-specific immune responses (i.e., at least 2 standard deviations above mean for negative controls for above assays). | Analysis.

CONTACTS AND LOCATIONS:
Locations (1):
- Saint Louis University - Center for Vaccine Development, St Louis, Missouri, United States